CLINICAL TRIAL: NCT07181590
Title: BaLloon-based PFA Ablation poST Approval Outcomes for PAF and PersAF
Acronym: BLAST-OFF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10608
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal AF; Atrial Arrhythmia; Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Pulsed Field Ablation; Persistent Field Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Volt PFA Catheter Sensor Enabled (SE) (Other): Patients diagnosed with drug refractory, symptomatic, recurrent, paroxysmal and persistent atrial fibrillation that will undergo a de novo ablation procedure with the Volt PFA Catheter.
  Interventions: Device: Pulsed Field Ablation

INTERVENTIONS:
Device: Pulsed Field Ablation — Pulsed Field Ablation using the Volt PFA System

SUMMARY:
This study is designed to obtain real-world clinical evidence on the safety and effectiveness of the Volt PFA System in various use cases, with a sub study designed to address additional clinical evidence needs in electrophysiology.

ELIGIBILITY:
Inclusion Criteria:

1. Documented symptomatic PAF or PersAF. Documentation requirements are as follows:

   Paroxysmal:
   * Physician's note indicating recurrent self-terminating AF AND
   * One electrocardiographically documented PAF episode within 12 months prior to enrollment.

   Persistent: Continuous AF sustained beyond 7 days and less than 1 year that is documented by
   * Physician's note, AND either
   * 24-hour Holter within 360 days prior to enrollment, showing continuous AF, OR
   * Two electrocardiograms (from any form of rhythm monitoring) showing continuous AF:

     * That are taken at least 7 days apart but less than 12 months apart
     * If electrograms are more than 12 months apart, there must be one or more Sinus Rhythm recordings in between or within 12 months prior to consent/enrollment
     * The most recent electrocardiogram must be within 180 days of enrollment.

   NOTE: Documented evidence of the AF episode must either be continuous AF on a 12-lead ECG or include at least 30 seconds of AF from another ECG device.
2. Plans to undergo a de novo ablation procedure with the Volt PFA Catheter due to symptomatic PAF or PersAF and is refractory, intolerant, or contraindicated to at least one Class I-IV AAD medication
3. At least 18 years of age
4. Able and willing to comply with all trial requirements including pre-procedure, post- procedure, and follow-up testing and requirements
5. Informed of the nature of the trial, agreed to its provisions, and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical trial site.

Exclusion Criteria

1. Arrhythmia due to reversible causes including thyroid disorders, acute alcohol intoxication, electrolyte imbalance, severe untreated sleep apnea, and other major surgical procedures in the preceding 90 days
2. Known presence of cardiac thrombus
3. Known Left ventricular ejection fraction < 35% as assessed with echocardiography within 360 days of index procedure
4. New York Heart Association (NYHA) class III or IV heart failure
5. Pregnant, nursing, or planning to become pregnant during the clinical investigation follow-up period
6. Patients who have had a ventriculotomy or atriotomy within the preceding 30 days of procedure
7. Myocardial infarction (MI), acute coronary syndrome, percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery within preceding 90 days
8. Unstable angina
9. Stroke or TIA (transient ischemic attack) within the last 90 days
10. Heart disease in which corrective surgery is anticipated within 180 days after procedure
11. History of blood clotting or bleeding abnormalities including thrombocytosis, thrombocytopenia, bleeding diathesis, or suspected anti-coagulant state
12. Contraindication to long term anti-thromboembolic therapy
13. Patient unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation
14. Previous left atrial surgical or left atrial catheter ablation procedure (including LAA closure device)
15. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2).
16. Previous tricuspid or mitral valve replacement or repair
17. Patients with prosthetic valves
18. Patients with a myxoma
19. Patients with an interatrial baffle or patch as the transseptal puncture could persist and produce an iatrogenic atrial shunt
20. Stent, constriction, or stenosis in a pulmonary vein
21. Rheumatic heart disease
22. Hypertrophic cardiomyopathy
23. Diagnosed with amyloidosis or atrial amyloidosis
24. Active systemic infection
25. Renal failure requiring dialysis
26. Severe pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
27. Presence of an implanted LAA closure device
28. Patient is currently participating in another clinical study that may confound the results of this of this post market evaluation; for example, enrolled in another study with an active treatment arm
29. Unlikely to survive the protocol follow up period of 12 months
30. Presence of other medical, anatomic, comorbid, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
31. Individuals without legal authority
32. Individuals unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects experiencing a device and/or procedure-related serious adverse event with onset within 7 days of any ablation procedure that uses Volt AF | 7 days
  Serious adverse events are defined as:
  * Atrio-esophageal fistula
  * Cardiac tamponade/perforation
  * Death
  * Heart block
  * Myocardial infarction
  * Pericarditis3
  * Phrenic nerve injury resulting in permanent diaphragmatic paralysis
  * Pulmonary Edema
  * Pulmonary vein stenosis1
  * Stroke
  * Thromboembolism
  * Transient ischemic attack
  * Vagal nerve injury/gastroparesis
  * Major vascular access complications4 / major bleeding events5
  * Device related cardiovascular and/or pulmonary adverse event that prolongs hospitalization for more than 48 hours (excluding hospitalization solely for arrhythmia recurrence or non-urgent cardioversion)
Long-term Effectiveness will be the proportion of subjects with freedom from documented AF/AFL/AT recurrence through 12-months. | During procedure
  Other situations in which subjects will be considered effectiveness endpoint failures include:
  * Cardioversion (electrical or pharmaceutical) for the treatment of AF/AFL/AT following the blanking period.
  * A second repeat procedure for ablation of AF recurrence within the 90-day blanking period
  * Any repeat ablation procedure in the left atrium (LA) for AF/AFL/AT following the 90-day blanking period
  * Any use of a new class I or III AAD for AF/AFL/AT after the 90-day blanking period
  * Any use of a class I or III AAD for AF/AFL/AT at a dose higher than the historical maximum dose for the subject after the blanking period.
Acute procedural effectiveness is defined as confirmation of entrance block in all targeted pulmonary veins | During procedure
  A secondary measure of confirmation to include any one of the following (the same method must be used for all pulmonary veins) :
  * A minimum 20-minute wait following initial confirmation of entrance block with a second confirmation of entrance block following the 20-minute wait; or
  * Exit block pacing maneuvers ; or
  * Isoproterenol or adenosine challenge

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Kammer, Study Director — Abbott Medical Devices
Locations (22):
- Ordensklinikum Linz Elisabethinen, Linz, Austria
- Belgium (2):
  - AZ Sint Jan, Bruges
  - UZ Brussel, Brussels
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - Hôpital Pitié Salpetrière, Paris
  - Hopital Haut Leveque, Pessac
  - Clinique Pasteur Toulouse, Toulouse
- Germany (4):
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen
  - Medizinische Einrichtungen der Universität zu Köln, Cologne
  - Asklepios Klinik St. Georg, Hamburg
  - TUM Klinikum - Deutsches Herzzentrum München, München
- Mater Private Hospital, Dublin, Ireland
- Italy (2):
  - Az. Osp.Universitaria Osp.Riuniti Umberto I-Lancisi-Salesi, Ancona
  - Centro Cardiologico Monzino, Milan
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - St. Antonius Ziekenhuis, Nieuwegein
- National Institute of Cardiology Warsaw, Warsaw, Poland
- ULS de Lisboa Ocidental, Lisbon, Portugal
- Spain (3):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia
- Karolinska University Hospital Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No